CLINICAL TRIAL: NCT07077967
Title: Impact of Artificial Lighting on Visual Acuity After Presbyopia Correction With an Extended Depth of Focus Intraocular Lens: Introduction of a Modified Luminous Efficiency Function V(λ)'
Brief Title: Luminous Efficiency Function V(λ)' of Patients That Underwent Pseudophakic Presbyopic Corrections With EDOF IOLs
Acronym: V(λ)'_EDOF
Status: Not yet recruiting | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: ES5/Th9/13-02-2025
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Presbyopia
Keywords: pseudophakic presbyopic correction; EDOF intraocular lens; light intensity; eye light transmittance; light efficiency function
MeSH Terms: conditions — Presbyopia | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients who underwent uneventful pseudophakic presbyopic correction with yellow filter extended depth-of-focus (EDOF) IOLs (Vivity or Vivity toric, Alcon Laboratories, Inc., Fort Worth, TX, USA)
  Interventions: Procedure: Phacoemulsification with EDOF IOLs
- Control group: Patients of similar age who underwent uneventful cataract surgery implanted with yellow filter monofocal or monofocal toric IOLs (SN60WF or SN6ATx, Alcon Laboratories, Inc., Fort Worth, TX, USA)

INTERVENTIONS:
Procedure: Phacoemulsification with EDOF IOLs — Uneventful pseudophakic presbyopic correction with EDOF IOLs
  Groups: Study group

SUMMARY:
Primary objective of this study is to introduce a modified luminous efficiency function that addresses the distinct total eye light transmittance of patients who underwent pseudophakic presbyopic correction with extended-depth of focus (EDOF) intraocular lenses (IOLs) implantations.

DETAILED DESCRIPTION:
Present study aims to identify in which degree EDOF IOLs modify eye light transmission and estimate the necessary task and environmental lighting adjustment in order to address lighting needs of patients following pseudophakic presbyopic corrections implanted with EDOF IOLs. Specifically, the aim of this study is to identify the minimum light intensity at which patients who underwent pseudophakic presbyopic correction with EDOF IOLs can reach their maximum visual acuity (measured when lights are at the 100% lighting level)

ELIGIBILITY:
Inclusion Criteria:

* age between 45 to 75 years

Exclusion Criteria:

* astigmatism >1.00 diopters
* glaucoma
* former incisional eye surgery
* corneal or fundus disease
* diabetes mellitus
* autoimmune diseases
* neurological or psychiatric diseases
* posterior capsule rupture or lens misalignment
* postoperative uncorrected distance visual acuity < 8/10.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Presbyopic patients who underwent pseudophakic presbyopic correction with EDOF intraocular lens implantation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Minimum Required Illuminance Level (MRIL) | 6 months postoperatively
  Minimum Required Illuminance Level (MRIL) (in lx) at which participants reach their optimal Uncorrected Distance Visual Acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Background] Labiris G, Panagiotopoulou EK, Taliantzis S, Perente A, Delibasis K, Doulos LT. Lighting Standards Revisited: Introduction of a Mathematical Model for the Assessment of the Impact of Illuminance on Visual Acuity. Clin Ophthalmol. 2021 Nov 28;15:4553-4564. doi: 10.2147/OPTH.S326139. eCollection 2021. PMID 34866900